CLINICAL TRIAL: NCT02483507
Title: Ultrasound-guided Peripheral Vascular Access: What Approaches in Paediatrics?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9420; 2013-A01587-38 (Registry Identifier: ID RCB)
Record Dates: First submitted 2015-06-15; First posted 2015-06-29 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2015-06

CONDITIONS: Pediatric Anesthesia; Comparison of 3 Peripheral Vascular Access
Keywords: Ultrasound guidance; Vascular access; Pediatric anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group T: transversal (Active Comparator): Implementation of the vascular catheter with transversal approach under ultrasound guidance
  Interventions: Other: Ultrasound-guided approach to peripheral vascular access
- Group L: longitudinal (Active Comparator): Implementation of the vascular catheter with longitudinal approach under ultrasound guidance
  Interventions: Other: Ultrasound-guided approach to peripheral vascular access
- Group O: oblique (Active Comparator): Implementation of the vascular catheter with oblique approach under ultrasound guidance
  Interventions: Other: Ultrasound-guided approach to peripheral vascular access

INTERVENTIONS:
Other: Ultrasound-guided approach to peripheral vascular access — the transversal approach is in short axis with an out of plane puncture, the longitudinal approach is in transversal axis with an in plane puncture, the oblique view approach is in obliques axis with an in plane puncture

SUMMARY:
Landmarks used to make a vascular puncture has long been based on the only knowledge of anatomy. This method assumes that the target vessel is in its expected position, permeable (non-thrombosed), and heavy enough to be catheterized. Any variations from these assumptions is likely to cause failures of puncture and complications. The development of ultrasound allowed to "see" the structures to achieve, whether before a puncture or in live for guiding the procedure. Visualization of vessels and adjacent structures has logically resulted in larger cases to a greater security of catheterization, improving the success rate, and decreasing complications. Several positions of the probe can be used to guide a puncture under ultrasound: the transversal approach in short axis, the long axis longitudinal approach and the oblique view approach.The aim of the study was to compare these three different ultrasound-guided approaches to peripheral vascular access in children. All children weighing less than 30 kg that should benefit from the introduction of an arterial catheter or central venous catheter introduced through a peripheral vein are eligible. Patients will be included after parent's and children's information and consent. The choice of the technique used (transverse, longitudinal or oblique approach) is determined by a randomization table.The puncture procedure is performed according to the usual protocols of the paediatric anesthesia unit of the investigators, under ultrasound guidance in a sterile manner. No time limit is required for the identification and implementation of the catheter. The position of the probe is dictated by the result of randomization and the Seldinger technique is used for the establishment of the catheter. Beyond two unsuccessful attempts, the procedure is considered as a failure. The anesthetist then uses the alternative technique of his choice. All anesthetists participating in this study exercised their main activity in the Montpellier University Hospital pediatric anesthesia unit. The laying of ultrasound-guided peripherally inserted central catheter and arterial catheter is part of the current activity of the unit.

ELIGIBILITY:
Inclusion Criteria:

1. Child requiring the implementation of a peripherally inserted central catheter or an arterial catheter.
2. Child whose general state corresponds to the Physical status score I - IV
3. Child whose weight is lower to 30 kg
4. Child whose parents will have given their informed consent.
5. Child affiliated to a national insurance scheme

Exclusion Criteria:

1. Child presenting a contraindication to the general anesthesia
2. Child whose weight is upper to 30 kg
3. Child whose parents did not give their informed consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2014-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Success rate | one hour
  The success of the procedure is defined by the success of the puncture to the first or the second attempt.

SECONDARY OUTCOMES:
The number of attempts | one hour
  the number of attempts is defined by the number of puncture performed
The duration of the puncture procedure | on hour
  the duration of the puncture procedure is defined for the puncture until objectivization of a blood reflux.
The operator satisfaction | one hour
  Level of satisfaction of the operators according to the technique used

CONTACTS AND LOCATIONS:
Overall Officials: Chrystelle CS SOLA, MD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Hôpital Lapeyronie - Département Anesthésie Réanimation A, Montpellier, France